CLINICAL TRIAL: NCT03402802
Title: Steroid Eyedrop Adherence After Trabeculectomy
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00160532
Record Dates: First submitted 2017-12-19; First posted 2018-01-18 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma; Adherence, Patient
Keywords: eye drop
MeSH Terms: conditions — Glaucoma; Patient Compliance | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: monitoring of adherence with medication — persons taking routine postoperative eye drops will have their frequency of drop taking monitored

SUMMARY:
The study will monitor how often persons use eye drops that are prescribed after glaucoma surgery and will compare the adherence with drop use to the success rate of the surgery.

DETAILED DESCRIPTION:
Trabeculectomy is the most common operation performed for all forms of glaucoma. The procedure depends upon appropriately modulated healing of the conjunctiva and sclera, a major component of which is delivery of frequent topical corticosteroid eye drops (prednisolone acetate 1%) by the patient, initially every 2 hours when awake for 1-2 weeks, then in tapering frequency over the 6 weeks after surgery. While the initial success of trabeculectomy at one year varies from 55-80% depending upon the criteria chosen to measure outcome, improvements in success would benefit hundreds of thousands of patients in the USA yearly. There is reasonable evidence that steroid drops benefit success, but there is essentially no data on how successfully patients remember to take the drops. In previous research, investigators have shown that glaucoma patients take only half to two-thirds of prescribed drops. An electronic monitoring device is now available that can fit the eye drop bottle used in steroid drops, accurately measuring the time and date of each drop taken. The investigators can further assess the accuracy with which each patient can deliver a drop from the bottle being monitored in a clinic session directly onto the eye's surface by observing their performance. The proposal's hypothesis is that the one year success rate of the procedure will be related to the adherence to steroid drop taking by patients. The outcome will have two important benefits. First, if adherence is less than ideal (which is very likely), then those with greater adherence will have more successful surgery, confirming that steroid treatment is effective. This has only been measured once, 30 years ago, at a time when trabeculectomy was being performed quite differently. If steroid treatment is not related to success, a change in preferred practice patterns is in order. If steroid treatment is related to success and adherence is variable, the investigation will have proven means to increase adherence through reminder systems, which have shown in past randomized clinical trial to be effective.

ELIGIBILITY:
Inclusion Criteria:

* Persons having glaucoma surgery

Exclusion Criteria:

* Persons not eligible for glaucoma surgery, including pregnant females persons allergic to standard postoperative eye drops

Ages: 21 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
adherence rate | 6 weeks
  frequency of taking eye drops

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Quigley, MD, Principal Investigator — Professor
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGlumphy EJ, Dosto NO, Johnson TV, Quigley HA. Electronically Monitored Corticosteroid Eye Drop Adherence after Trabeculectomy Compared to Surgical Success. Ophthalmol Glaucoma. 2022 Jul-Aug;5(4):379-387. doi: 10.1016/j.ogla.2021.12.007. Epub 2022 Jan 4. PMID 34995818